CLINICAL TRIAL: NCT06516263
Title: A Randomised Control Clinical Trial Investigating the Effect of L-PRF on Implant Stability and Marginal Bone Levels.
Brief Title: Effect of L-PRF on Implant Stability and Marginal Bone Levels.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dublin Dental University Hospital (Other)
Responsible Party: Principal Investigator, Daniel Merrick, Principal Investigator, Dublin Dental University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DublinDental
Record Dates: First submitted 2024-07-12; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Dental Implant; Implant Stability; Marginal Bone Levels; L-PRF
MeSH Terms: interventions — Leukocyte Count

STUDY DESIGN:
Intervention Model Description: This is a parallel arm, randomised control clinical Trial (RCT) on a cohort of Dublin Dental University Hospital patients who are having dental implants placed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The effect of Leukocyte and platelet rich fibrin on Implant Stability and Marginal Bone Levels. (Experimental): Standard Implant placement with Leukocyte and platelet rich fibrin
  Interventions: Procedure: Leukocyte and platelet rich fibrin
- The Effect of standard implant placement on implant Stability and Marginal Bone Levels. (Placebo Comparator): standard implant placement
  Interventions: Procedure: Standard implant placement

INTERVENTIONS:
Procedure: Leukocyte and platelet rich fibrin — Formation of an Leukocyte and platelet rich fibrin clot and placement into the osteotomy site prior to implant placement
  Arms: The effect of Leukocyte and platelet rich fibrin on Implant Stability and Marginal Bone Levels.
Procedure: Standard implant placement — Standard implant placement without Leukocyte and platelet rich fibrin
  Arms: The Effect of standard implant placement on implant Stability and Marginal Bone Levels.

SUMMARY:
Osseointegration refers to the formation of a structure and functional bone-to-bone interface, without the interposition of soft tissue. Successful osseointegration is imperative to implant success and relies on a number of factors including implant design, material, surface and finish the bone status, surgical technique and implant loading conditions. Primary implant stability is the bio-mechanical stability achieved for implants at the time of placement and is achieved through micromovements of the implant. Following healing of the osteotomy site and formation of new bone a biological fixation of the implant to bone results and is referred to as secondary implant stability. Such as with osseointegration, there are several factors that affect primary implant stability including insertion torque, implant design, density of bone and surgical technique. To achieve future implant osseointegration, primary stability must first be accomplished.

Leukocyte and platelet rich fibrin (L-PRF) is formed by centrifuging venous blood using an IntraSpin® machine (U.S Food and Drug Administration approved and CE marked for in-vivo use) at 2700 revolutions per minute for 12 minutes. Following removal from the L-PRF tubes the fibrin clot is separated from the red blood cell clot. The fibrin clot is then transferred to the PRF box and the Xpression™ tray is placed over the fibrin clot and after 5 minutes the L-PRF membrane is ready for use.

During the traditional implant placement there is an osteotomy cut in practical terms is a controlled fracture of the bone resulting in rupture of local blood vessels which almost immediately sparks a cascade of healing including hemostasis, inflammation and proliferation of cells and tissue maturation. Our study will include Leukocyte platelet rich fibrin surrounding the implant at the osteotomy site which is a robust fibrin mesh which provides a progressive release of growth factors improving angiogenesis, osteoblastic proliferation, and cell differentiation. L-PRF utilization during implant placement attempts to expedite the process by delivering growth factors to the surface of the implant and surrounding bone promoting the healing process. Experimental research has shown that delivery of molecules or growth factors to an implants surface may increase osteoblast activity and improve functional integration of the implant.

Pre-clinical tests have shown that the utilization of platelet growth factors improve wound healing, proliferation of cells and implant osseointegration in animal models. Further pre-clinical studies have shown that L-PRF increased the rate and amount of new bone formation in rabbits.

Limited human tests in small populations not including the mandible have shown positive outcomes with improvement in implant stability when L-PRF was utilized during implant placement. High quality clinical evidence on this topic is limited and must be improved to allow clinicians to make evidence-based decisions on L-PRF utilization.

The proposed study will be a randomized control trial comparing the use of L-PRF in implant placement versus conventional implant placement. Considering the extra step of phlebotomy and time for centrifuging of the blood samples the literature must show a clinical benefit if this technique is to be utilized into the future. This study aims to add to available clinical evidence and address some of the limitations in current evidence to aid clinicians to make evidence-based decisions on whether to utilize LPRF to improve implant stability and hence earlier loading of implants.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

Patient Level

* Male or Female, 18 years old or over
* Capacity to provide informed consent
* Willing to comply with study appointment schedule Willing to maintain a diary of symptoms
* Planned for provision of dental implant(s) at Dublin Dental University Hospital Site Level
* Location: maxilla and mandible
* Sufficient bone volume for implant placement without the need for bone graft/augmentation; alveolar ridge of minimum 6mm width for standard implants (implant diameter 4mm) and of minimum 7mm for wider implants (implant diameter 5mm)

Exclusion Criteria:

* Patient Level
* Plaque score >20%
* Bleeding score >20%
* Tobacco smoking
* Uncontrolled systemic disease
* Use of systemic medications with an expected impact on bone healing (e.g. bisphosphonates)
* Pregnancy or lactation
* lack of capacity to give informed consent
* Previous radiation to the head and/or neck Site Level
* Insufficient bone volume for implant placement, requiring bone graft/augmentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Implant stability quotient | baseline, 3 months and 4-6 months
  taken as Implant stability quotient value with an OSTELL device

SECONDARY OUTCOMES:
Pain levels | After anaesthetic has worn off, 24 hours and 1 week
  Pain levels recorded on Visual Analogue Scale
Clinical Marginal bone levels | Measured clinically at baseline and 3 months after implant placement at second stage surgery
  measure of implant to crest of bone
Radiographic marginal bone levels | at baseline 3 months and 4-6 months following implant placement
  measurement of crest of bone to implant on radiograph

CONTACTS AND LOCATIONS:
Locations (1):
- Dublin Dental University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
During collection the pseudo anonymized/coded data will be saved separately from the patients' dental charts on a password protected Dublin Dental University Hospital (DDUH) computer. The information will remain confidential from other DDUH health care staff, who can view patients' records.
  b) Following collection of the data, they will be processed to become anonymous (The identification key will be deleted). All anonymized data will be stored on a password protected DDUH computer with access granted only to the investigator and supervisor.
  c) It is not anticipated that there will be any hardcopy records arising from this study d) All data will be securely retained for 5 years after their analysis according to best practice regulations. - Five years after their original analysis, all data will be destroyed. All electronic data will be permanently deleted.